CLINICAL TRIAL: NCT04142970
Title: A Clinical Study Comparatively Evaluating the Pharmacokinetics, Pharmacodynamics and Safety of Intravenous Administration of HSK3486 Injectable Emulsion in Patients With Chronic Renal Impairment and Subjects With Normal Renal Functions
Brief Title: Safety and Pharmacokinetics/Pharmacodynamics of HSK3486 in Patients With Impairment Renal Functions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: HSK3486-106
Record Dates: First submitted 2019-10-24; First posted 2019-10-29 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Chronic Renal Impairment
Keywords: Mild renal impairment; Moderate renal impairment
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — HSK3486

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild renal impairment (Active Comparator): Mild renal impairment (eGFR: 60-89 mL/min/1.73 m^2)
  Interventions: Drug: HSK3486
- Moderate renal impairment (Active Comparator): Moderate renal impairment (eGFR: 30-59 mL/min/1.73 m^2)
  Interventions: Drug: HSK3486
- Subjects with normal renal functions (Active Comparator): Subjects with normal renal functions (eGFR: ≥ 90 mL/min/1.73 m^2)
  Interventions: Drug: HSK3486

INTERVENTIONS:
Drug: HSK3486 — HSK3486，Initially 0.4 mg/kg was administered as a 1 minute bolus, followed immediately by a constant infusion dose of 0.4 mg/kg/h administered as a 30 minute infusion via infusion pump.

SUMMARY:
A Clinical Study Comparatively Evaluating the Pharmacokinetics, Pharmacodynamics and Safety of Intravenous Administration of HSK3486 Injectable Emulsion in Patients with Chronic Renal Impairment and Subjects with Normal Renal Functions

DETAILED DESCRIPTION:
This is a single-center, open-label, non-randomized, parallel-controlled Phase I clinical study carried out in subjects with varying degrees (mild or moderate) of renal impairment, and age-, weight-, and gender-matched subjects with normal renal functions.

ELIGIBILITY:
Subject Inclusion Criteria (Must Meet All of the Following Criteria):

Inclusion Criteria:

1. Males or females with full capacity for civil conduct, aged ≥ 18 and < 65 years old;
2. Weighing ≥ 45 kg, and with a body mass index (BMI) of ≥ 18 and ≤ 28 kg/ m^2(BMI = weight (kg)/height2 ( m^2));
3. For matched subjects with normal renal functions: physical examination, laboratory tests (blood routine, blood biochemistry, urine routine, urinary albumin/creatinine ratio, creatine kinase (CK) and coagulation function), and 12-lead ECG, etc. should be normal or abnormal without clinical significance as determined by the investigator;
4. No potential difficult airway (modified Mallampati score of Grade I to II);
5. For matched subjects with normal renal functions: no history of major organ primary diseases, such as liver, kidneys, digestive tract, blood, and metabolic diseases; no history of malignant hyperthermia and other genetic conditions; no history of mental/neurological diseases; no history of epilepsy; no contraindications for deep sedation/general anesthesia; no clinically significant history of anesthesia accidents;
6. Subjects must understand the procedures and methods of this study, and be willing to signing the informed consent form and to complete the trial in strict accordance with clinical trial protocol;

   Patients with Renal Impairment Must Also Meet the Following Criteria:
7. The estimated glomerular filtration rate (eGFR) of the subjects in corresponding groups meets the criteria for mild to moderate renal impairment in the staging of renal functions, i.e., mild renal impairment: 60-89 mL/min/1.73 m^2; moderate renal impairment: 30-59 mL/min/1.73 m^2; subjects with normal renal functions: ≥ 90 mL/min/1.73 m^2;
8. For subjects with renal impairment, their laboratory test results (coagulation function, blood routine, urinary albumin/creatinine ratio, creatine kinase (CK), blood biochemistry, and urine routine) should be judged by the investigators as clinically stable and consistent with the severity of their renal impairment. In addition, their albumin should be > 35 g/L and hemoglobin should be > 110 g/L;

Exclusion Criteria( those who meet any one of the followings are ineligible):

1. Known sensitivity to excipients in HSK3486 injectable emulsion (soybean oil, glycerin, triglyceride, egg lecithin, sodium oleate and sodium hydroxide); history of drug allergies (including other anesthetics);
2. Received any one of the following medications or treatments prior to screening/enrollment:

   History of drug abuse or any signs of long-term use of benzodiazepines (such as insomnia, anxiety, spasms) within 3 months prior to screening; Participated in clinical trials involving any medications or medical devices within 3 months prior to screening, or subjects who have participated in 3 or more drug clinical trials within the past year; Serious infection, trauma, or major surgery within 4 weeks before screening; or acute disease with clinical significance (determined by the investigators) within 2 weeks before screening, including GI diseases or infections (such as respiratory tract or CNS infections); In receipt of propofol, other sedatives/anesthetics and/or opioid analgesics or compounds containing analgesics within 72 hrs prior to baseline; Used potent inhibitors of CYP enzyme within 7 days prior to enrollment, or used moderate/low potency inhibitors of CYP enzyme within 3 days prior to enrollment;
3. History or evidence of any one of the following diseases prior to screening/enrollment:

   History of cardiovascular diseases such as: uncontrolled hypertension [SBP ≥ 170 mmHg and/or DBP ≥ 105 without antihypertensive treatment, or SBP > 160 mmHg and/or DBP > 100 mmHg despite antihypertensive treatment], postural hypotension, severe arrhythmia, heart failure, Adams-Stokes syndrome, unstable angina, myocardial infarction within 6 months before screening, history of tachycardia/bradycardia requiring medication, II-III degree atrioventricular block (excluding patients with pacemakers) or QTcF interval ≥ 450 ms (Fridericia's correction formula); Respiratory insufficiency, history of obstructive pulmonary disease, history of asthma, sleep apnea; history of failed tracheal intubation; history of bronchospasm requiring treatment within 3 months prior to screening; acute respiratory infection, and with obvious symptoms such as fever, wheezing, nasal congestion or cough within 1 week prior to baseline; History of gastrointestinal diseases: History of gastrointestinal retention, moderate and above active bleeding (GUSTO bleeding classification), gastroesophageal reflux that may lead to aspiration; [Note: GUSTO bleeding classification is: heavy or life-threatening bleeding (intracranial hemorrhage or bleeding that causes hemodynamic compromise and requires intervention), moderate bleeding (requires blood transfusion but does not cause hemodynamic compromise), minor bleeding (does not meet the criteria for either severe or moderate bleeding)]; History of cerebrovascular diseases: history of craniocerebral injury, possible convulsions, intracranial hypertension, cerebral aneurysm, or cerebrovascular accident; History of mental illness: schizophrenia, mania, chronic use of antipsychotics, or cognitive impairment;
4. Positive test for either HBsAg, HCV, HIV, or syphilis;
5. History of alcohol abuse within 3 months prior to screening, alcohol abuse defined as average of > 2 units of alcohol per day (1 unit = 360 mL beer or 45 mL liquor with 40% alcohol or 150 mL wine), or positive alcohol breath test results at baseline;
6. Smoke more than 5 cigarettes per day and a total of more than 60 cigarettes within 3 months prior to screening;
7. Blood donation or blood loss ≥ 200 mL within 30 days prior to screening; plasma donation or plasma exchange within 7 days prior to screening;
8. Subjects who have consumed any beverages or foods containing alcohol, grapefruit juice or methylxanthine (such as coffee, tea, cola, chocolate, and functional drinks), participated in strenuous physical activities and other factors that may affect drug absorption, distribution, metabolism, and excretion within 2 days prior to baseline; subjects who are unable to fast for 8 hrs before dose administration;
9. Subjects expected to have surgery or hospitalization during the trial;
10. Subjects unsuitable for arterial blood collection, such as subjects who have positive Allen's test results;
11. Other than the disease diagnosed as renal impairment, patients with acute illnesses in any other organ, as well as those with chronic conditions that may affect the in vivo process of the investigational drug (e.g., chronic hepatitis, hepatic insufficiency, etc.);
12. Patients with autoimmune nephropathy, obstructive nephropathy, history of kidney transplantation, and an ongoing dialysis treatment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | -30 minutes before administration until 24 hours post administration on day 1
  Cmax（a measure of the body's exposure to HSK3486）will be compared between normal renal function patients and mild or moderate chronic renal impairment patients .
Area under the concentration-time curve（AUC） | -30 minutes before administration until 24 hours post administration on day 1
  AUC（a measure of the body's exposure to HSK3486）will be compared between normal renal function patients and mild or moderate chronic renal impairment patients .

SECONDARY OUTCOMES:
MOAA/S(modified observer's assessment of alert /sedation) | -5 minutes before administration until 1 hours post administration on day 1
Bispectral index(BIS) | -5 minutes before administration until 1 hours post administration on day 1
Tmax | -30 minutes before administration until 24 hours post administration on day 1
  time to peak observed
Total clearance | -30 minutes before administration until 24 hours post administration on day 1
Volume of distribution | -30 minutes before administration until 24 hours post administration on day 1
blood pressure（systolic, diastolic and mean arterial pressure） | from the screening to 3 days post-dose
  safety endpoits

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Tao J, Liu S, Zhao YY, Qi L, Yan P, Wu N, Liu X, Liu D, Tian X. Pharmacokinetics, pharmacodynamics, and safety of ciprofol emulsion in Chinese subjects with normal or impaired renal function. Front Pharmacol. 2023 Nov 23;14:1260599. doi: 10.3389/fphar.2023.1260599. eCollection 2023. PMID 38074142